CLINICAL TRIAL: NCT06936852
Title: Ultrasound Guided Serratus Posterior Superior Intercostal Plane Block Versus Pectoral Nerve (PECS II) Block For Pain Control In Breast Surgeries: A Randomized Controlled Trial
Brief Title: Ultrasound Guided Serratus Posterior Superior Intercostal Plane Versus PECS II Block In Breast Surgeries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Wahed Ali, lecturer at Anesthesia & Surgical ICU and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1097/2/25
Record Dates: First submitted 2025-03-30; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
Keywords: serratus posterior superior; pecs; breast surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIP Group (Active Comparator): Under complete aseptic technique, a high frequency linear probe will be placed adjacent to upper medial part of scapula to visualize the second and third ribs. The needle will be introduced with in plane approach, from caudal to cranial and 30 ml of 0.25% bupivacaine will be injected in the fascial plane between serratus posterior superior and intercostal muscles at the level of second and third ribs.
  Interventions: Procedure: Serratus posterior superior intercostal plane block
- PECS II group (Active Comparator): Under complete aseptic technique, a high frequency linear probe will be placed in the infraclavicular region, angulated and directed laterally towards the axilla to visualize the third and fourth ribs with pectoralis major, minor and serratus anterior muscles from superficial to deep. The needle will be introduced with in plane approach from medial to lateral, 10 ml of 0.25% bupivacaine will be injected in the fascial plane between pectoralis major and pectoralis minor then the needle will be further introduced to the fascial plane between pectoralis minor and serratus anterior muscles with injection of 20 ml of 0.25% bupivacaine.
  Interventions: Procedure: PECS II block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block — Under complete aseptic technique, a high frequency linear probe will be placed adjacent to upper medial part of scapula to visualize the second and third ribs. The needle will be introduced with in plane approach, from caudal to cranial and 30 ml of 0.25% bupivacaine will be injected in the fascial plane between serratus posterior superior and intercostal muscles at the level of second and third ribs.
  Arms: SPSIP Group
Procedure: PECS II block — . Under complete aseptic technique, a high frequency linear probe will be placed in the infraclavicular region, angulated and directed laterally towards the axilla to visualize the third and fourth ribs with pectoralis major, minor and serratus anterior muscles from superficial to deep. The needle will be introduced with in plane approach from medial to lateral, 10 ml of 0.25% bupivacaine will be injected in the fascial plane between pectoralis major and pectoralis minor then the needle will be further introduced to the fascial plane between pectoralis minor and serratus anterior muscles with injection of 20 ml of 0.25% bupivacaine.
  Arms: PECS II group

SUMMARY:
The aim of the study is to compare the analgesic effect of ultrasound guided serratus posterior superior intercostal plane (SPSIP) block and pectoral nerve (PECS II) block in different breast surgeries.

DETAILED DESCRIPTION:
All patients will be seen in the anesthesia clinic, optimization of general condition and all required investigations will be done before surgery. Patients will be premedicated with 1.5 mg midazolam and 4 mg granisetron. Standard basic monitoring will be applied to all patients then after adequate preoxygenation, induction of general anesthesia will be done through wide bore cannula using 1 mic/kg fentanyl, 1-2 mg/kg titration of propofol, 0.5mg/kg atracurium. Patients were mechanically ventilated using volume-controlled ventilation (VCV) with adjustment of end tidal carbon dioxide (ETCO2) to be 32-35 mmHg, 50% inspired oxygen in air and sevoflurane concentration to be 1MAC. The patients will receive either block before skin incision that will be done 20 minutes after the block. 0.5 mic/kg fentanyl will be injected when heart rate or blood pressure increases more than 20% of baseline. By the end of the surgery, 1gm paracetamol will be administered with fully reversal of muscle relaxants at the end of the surgery.

SPSIP group After induction of anesthesia, patients will be placed in lateral decubitus position, the affected arm will be adducted and medially rotated. Under complete aseptic technique, a high frequency linear probe will be placed adjacent to upper medial part of scapula to visualize the second and third ribs. The structures from superficial to deep are skin, subcutaneous, trapezius, rhomboid, serratus posterior superior and intercostal muscles. The needle will be introduced with in plane approach, from caudal to cranial and 30 ml of 0.25% bupivacaine will be injected in the fascial plane between serratus posterior superior and intercostal muscles at the level of second and third ribs.

PECS II group With the patient in supine position, the ipsilateral upper arm will be abducted and externally rotated. Under complete aseptic technique, a high frequency linear probe will be placed in the infraclavicular region, angulated and directed laterally towards the axilla to visualize the third and fourth ribs with pectoralis major, minor and serratus anterior muscles from superficial to deep. The needle will be introduced with in plane approach from medial to lateral, 10 ml of 0.25% bupivacaine will be injected in the fascial plane between pectoralis major and pectoralis minor then the needle will be further introduced to the fascial plane between pectoralis minor and serratus anterior muscles with injection of 20 ml of 0.25% bupivacaine.

After extubation, the patients will be transferred to PACU (Post-Anesthesia Care Unit) for monitoring. Numerical rating scale (NRS) will be used for pain assessment while 0 is no pain and 10 is severe agonizing pain. Patients will be given a rescue analgesia of 0.05 mg / kg morphine if NRS ≥ 4 and repeated if needed. Intravenous 1 gm paracetamol every 8 h and 30 mg ketorolac (if not contraindicated) every 12 h will be given regularly.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 70 years, both male and female.
* American Society of Anesthesiologists (ASA) Physical Status Classification System I-II.

Exclusion Criteria:

* Any patient refuses to participate.
* Bleeding or coagulation disorders, hepatic dysfunction, psychiatric diseases.
* Chronic opioid use.
* History of allergy to local anesthetics.
* Infection at the needle entry point will be excluded.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | first postoperative 24 hour
  Total morphine consumption in first postoperative twenty four hour

SECONDARY OUTCOMES:
NRS when reaching recovery room arrival, after 2 hour, 6 hour, 12 hour, 18 hour, 24 hour | when reaching recovery room (average 10 minutes after surgery), after two, six, twelve, eighteen, twenty four hour
  NRS when reaching recovery room, after 2 hour, 6 hour, 12 hour, 18 hour, 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Select, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Gundogdu O, Avci O, Balci F, Tekcan MN, Kol YC. Efficacy of Serratus Posterior Superior Intercostal Plane Block on Postoperative Pain and Total Analgesic Consumption in Patients Undergoing Reduction Mammoplasty Surgery: An Evidence Based Report. J Coll Physicians Surg Pak. 2024 Mar;34(3):348-350. doi: 10.29271/jcpsp.2024.03.348. PMID 38462873